CLINICAL TRIAL: NCT03395431
Title: The Feasibility of Fingerprick Autologous Blood (FAB) As a Novel Treatment for Severe Dry Eye Disease (DED)
Brief Title: Fingerprick Autologous Blood (FAB) in Severe Dry Eye Disease (DED)
Acronym: FAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bedford Hospital NHS Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 233813
Record Dates: First submitted 2017-11-02; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-11

CONDITIONS: Dry Eye Syndromes
Keywords: Autologuous serum; dry eyes disease; fingerprick blood
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A single blind parallel group randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAB group (Active Comparator): Arm A - Finger prick autologous blood (FAB) plus conventional treatment The patients will use FAB alongside conventional therapy as recommended by their treating ophthalmologist. A fingertip of the hand will be wiped with an alcohol steret and self-pricked using a standard diabetic lancet. The drop of blood is produced as normal and applied to the lower fornix of the affected eye(s) with the lower lid pulled down slightly by the patient. The blood will be applied 4 times a day. A fresh finger should be used for each eye. FAB should be applied at least 15 minutes after any artificial tears and no other drops applied for at least half an hour afterwards
  Interventions: Other: Fingerprick autologuos blood (FAB)
- Control group (No Intervention): Arm B - Conventional treatment only The patients will use conventional therapy (artificial tears, cyclosporin drops and punctal plugs/cautery) as recommended by their treating ophthalmologist

INTERVENTIONS:
Other: Fingerprick autologuos blood (FAB) — Intervention involves the instillation of whole blood obtained from the prick of a clean finger 4 times a day.
  Other Names: FAB
  Arms: FAB group

SUMMARY:
Dry eye disease (DED) is an umbrella term encompassing a range of diseases estimated to affect 14% of all adults aged 48 to 91. If left untreated, DED can lead to severe reduction in the quality of life of the sufferer. It can also cause loss of vision, pain in response to light, painful recurring stabbing sensations, and the feeling of grit in the affected eye(s). No curative agents for DED exist. Available conventional treatment options for DED such as artificial tears often only alleviate symptoms, have limited effectiveness, and in most cases patients may fail to respond; although the exact rate of treatment failure is unavailable in the published literature. Crudely, human tears with its vast constituents is essentially filtered blood and as such is an obvious source for a "tear mimic" containing the substances of tears. Blood, and several blood derived products, including autologous serum, have been studied as tear substitute candidates. This study proposes to test the use of finger prick autologous blood (FAB) technique in which whole blood is applied to the eye from a cleaned finger.

DETAILED DESCRIPTION:
Autologous serum (AS) eye drops have been found in uncontrolled trials to be beneficial in DED patient by improving the ocular surface and reducing symptoms. Obtaining autologous serum requires frequent drawing of blood from the patient- a feature that excludes patients with anaemia or heart failure from using AS. Furthermore it also appears that 100% autologous serum is more beneficial than 50% serum and requires larger volumes of blood and/or more frequent venesection. Patients using AS also require access to a fridge as the product needs to be stored at low temperatures; a factor that is likely to be inconvenient for patients. In addition, AS is obtained by processing clotted blood which is often too expensive for the health service to consistently purchase, given the initial cost of £1653.56 and subsequent three-monthly cost of £1131.27 per patient.

The relatively high cost represents the biggest hurdle in the use of AS and is often the reason for delay or inaccessibility in starting treatment for DED using AS. However, we propose that finger prick autologous blood may be a simpler, cost-effective and possibly more acceptable method for treating dry eye disease. For this reason, this study proposes to test the use of finger prick autologous blood (FAB) technique in which whole blood is applied to the eye from a cleaned finger.

The proposing team have completed an exploratory study on the use of finger-prick autologous blood (FAB) for persistent epithelial defects and severe dry eye disease and preliminary results indicate improvement with no adverse events reported. The exploratory study included 16 patients with a diagnosis of severe to moderate dry eye syndrome and used the FAB method for treatment. The findings of the study demonstrated mean improvements in visual acuity, Oxford corneal staining grade, tear breakup time, Schirmer's test and dry eye disease questionnaire score. The response rate from participants was good with only a single patient who met the inclusion criteria not wishing to participate in the trial on the advice of their general practitioner. Both the amount of staining (indicating inflammation and ocular surface damage) and their DED questionnaire scores (indicating severity of their symptoms and impact on quality of life) showed mean improvement which reached statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Severe symptomatic dry eye disease diagnosed by: Ocular surface disease index (OSDI) score of greater than 33; OR Oxford Corneal Staining grade 2 or greater; OR Schirmer's without anaesthesia <5mm at 5 minutes
* Patients on artificial tears and/or lubricating drops/gel two or more times a day
* Patient able to give consent
* Patients able and willing complete the quality of life (QoL) questionnaires required for the study

Exclusion Criteria:

* Fear of needles
* Unable or not willing to carry out repeat finger pricks
* Patients with infected finger/s or systemic infection or on systemic antibiotics for infection.
* Patients with active ocular infection, active immunological corneal melt, or recurrent corneal erosion.
* Pregnant or breast feeding women
* Previous use of FAB treatment (e.g. from exploratory study)
* Systemic illness causing immune system deficiency
* Graft versus host disease
* Previous use of autologous serum within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited into the study within the specified time frame | 12 months
  This will involve specifically assessing the number of eligible patient in study population consented and randomized.
Number of patients who adhere to trial protocol | 12months
  Measured by self-reported adherence to trial protocol

SECONDARY OUTCOMES:
Reduction in corneal inflammation as indicated by staining on front of the eye | 3 months
  Assessed using the Oxford Corneal Staining Guide graded on a scale from 0 to 5 in order of increasing severity
Patient pain and symptoms scores | 3 months
  This will be assessed by Ocular Surface Disease Index (OSDI) score assessed on a scale of 0 to 100 with higher score representing severity
Improvement in objective signs of dry eye disease as indicated by visual acuity | 3 months
  This will be assessed using the Snellen chart
Willingness for patients to be randomised and acceptability of the intervention | 3 months
  This will be assessed by structured qualitative interviews
Impact on patients' quality of life | 3 months
  This will be assessed by EQ-5D-5L score with higher scores indicating improvement in quality of life
Cost to the NHS and patient | 3 months
  This will be assessed by use of additional NHS services and privately purchased over the counter treatments related to dry eyes disease
Intraocular pressure (IOT) | 3 months
  Intraocular pressure will be measured to assessed safety of the intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poon AC, Geerling G, Dart JK, Fraenkel GE, Daniels JT. Autologous serum eyedrops for dry eyes and epithelial defects: clinical and in vitro toxicity studies. Br J Ophthalmol. 2001 Oct;85(10):1188-97. doi: 10.1136/bjo.85.10.1188. PMID 11567963
- [Background] Tsubota K, Goto E, Fujita H, Ono M, Inoue H, Saito I, Shimmura S. Treatment of dry eye by autologous serum application in Sjogren's syndrome. Br J Ophthalmol. 1999 Apr;83(4):390-5. doi: 10.1136/bjo.83.4.390. PMID 10434857
- [Background] Fox RI, Chan R, Michelson JB, Belmont JB, Michelson PE. Beneficial effect of artificial tears made with autologous serum in patients with keratoconjunctivitis sicca. Arthritis Rheum. 1984 Apr;27(4):459-61. doi: 10.1002/art.1780270415. No abstract available. PMID 6712760
- [Background] Than J, Balal S, Wawrzynski J, Nesaratnam N, Saleh GM, Moore J, Patel A, Shah S, Sharma B, Kumar B, Smith J, Sharma A. Fingerprick autologous blood: a novel treatment for dry eye syndrome. Eye (Lond). 2017 Dec;31(12):1655-1663. doi: 10.1038/eye.2017.118. Epub 2017 Jun 16. PMID 28622325
- [Derived] Balal S, Udoh A, Pappas Y, Cook E, Barton G, Hassan A, Hayden K, Bourne RRA, Ahmad S, Pardhan S, Harrison M, Sharma B, Wasil M, Sharma A. The feasibility of finger prick autologous blood (FAB) as a novel treatment for severe dry eye disease (DED): protocol for a randomised controlled trial. BMJ Open. 2018 Oct 31;8(10):e026770. doi: 10.1136/bmjopen-2018-026770. PMID 30385451